CLINICAL TRIAL: NCT03785119
Title: Improvement of in Vitro Fertilization Implantation by Soluble CD146 Dose in Embryonic Culture Environment : Multicenter Prospective Study
Brief Title: Improvement of in Vitro Fertilization Implantation by Soluble CD146 Dose in Embryonic Culture Environment
Acronym: AMIFIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-20
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: in Vitro Fertilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard strategy: According to embryo quality (morphologic criteria)
- Experimental strategy: Association of embryo quality and sCD146 rate

SUMMARY:
The study of implantation potential of the embryo stay a priority in In Vitro Fertilization (IVF). Indeed, the selection of embryos to transfer is actually based in routine check on morphologic criteria, approved by literature but not perfect. Implantation's markers identification, allowing to choose the embryo(s) to transfer and then decrease pregnancy failure, represent a major issue in IVF, not any biomarker being approved yet.

Among factors regulating embryonic implantation, investigators have recently proposed soluble CD146, coming from proteolytic cleavage of the CD146 membrane, angiogenic bond molecule.

In a monocentric study about 222 transferred embryos at the end of IVF try, investigators showed that the sCD146 dose in the embryonic culture environment reflected the implantation ability of embryo, a high rate showing a low implantation potential and this independently of the embryonic quality. A multicentric prospective study is now required to confirm the utility of this dosage in clinical practice.

Primary objective : Compared 2 frozen embryo transfer (FET) strategies in terms of implantation efficiency, according to choice method of embryo to be transferred :

* Group A : Standard strategy : Depending on embryonic quality according to criteria currently selected.
* Group B : Experimental strategy : Association of embryonic quality according to criteria currently selected and of sCD146 rate.

Expected Results :

* Demonstrate a beginning pregnancy test significantly superior in Group B compared to Group A.
* Confirmed that sCD146 is an independent biomarker of morphologic embryonic quality (actual selection criteria) and represent a complementary criteria to choose embryos to transfer.

Methodology :

- Multicentric prospective study with 2 groups of Frozen Embryo Transfer (FET); The calculation of the number of staff required includes 151 couples per group.

For this will be include for 24 months, couples benefiting of freezing at least one of the two embryos and transfer of only one FET.

* Test the same day of environment freezing where frozen embryos were cultivated. sCD146 dosage by ELISA technic (Enzyme Linked ImmunoSorbent Assay) in thus culture environment before FET.
* Implantation potential analyze of each transfer embryo (FET) according to sCD146 rate.
* Following of the FET future(pregnancy, childbirth) : maximum 9 months after attempt to each included couple.

ELIGIBILITY:
Pre Inclusion Criteria:

* Women aged [18;42] years
* Men aged > 18 years
* Trying an IVF with :
* Frozen supernumerary embryo after fresh embryo transfer realised at the end of the try or frozen embryo (frozen all), without immediately transfer possibility (ovulation hyperstimulation context/ hyperprogesteronemia for example)
* Freezing at least 2 embryos frozen separately (1/vial)
* Whatever attempt rank
* Whatever MAP (Medically Assisted Procreation) technics (IVF/ICSI)
* Potential transfer of one frozen embryo
* Volunteer couples to participate at the study, received informations about this protocol and giving both their non opposition

Inclusion Criteria:

- FET realization in the selected population

Exclusion Criteria:

* Refusal to participate at the study of at least one member of the couple
* Inclusion realized for a previous attempt
* IVF try with a third-party
* IVF try without embryo freezing
* Freezing only one embryo
* Non separately freezing of embryos (2/vial)
* Female patients <18 years and >42 years
* Male patients <18 years

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples benefiting of at least one of the two embryos and a transfer of one frozen embryo (FET)
Sampling Method: Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Beginner pregnancy rate at 1st transfer (%) | 0 to 9 months after FET
  Corresponds to number of defined pregnancy by plasmatic quantity of hCG (human chorionic gonadotropin) >100 UI/l 15 days after FET/number of FET.

SECONDARY OUTCOMES:
Beginner pregnancy rate at 2nd or 3rd transfer | 0 to 9 months after FET
  Corresponds to number of defined pregnancy by plasmatic quantity of hCG >100 UI/l 15 days after FET/number of FET.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service de Biologie de la Reproduction, Marseille, France